CLINICAL TRIAL: NCT07177989
Title: Combined Effects of Alternate Nostril Breathing and Aerobic Interval Training on Blood Pressure and Heart Rate Products in Patients With Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/92
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension (HTN)
Keywords: hypertension; intensity interval training; nostril breathing; heart rate; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group (Group B), will receive alternative nostril breathing along with aerobic interval training and the other group group B) will receive only aerobic interval training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Group B) (Experimental): Patients in this group will perform alternative nostril breathing along with aerobic interval training.
  A protocol of total 5 weeks. Three sessions per week on alternate days will be done under the supervision of physiotherapist.
  All outcome measurements would be performed first at baseline and terminal after the 5 weeks intervention period
  Interventions: Other: Experimental Group
- Interventional group (Group A) (Active Comparator): Patients in tis group will perform aerobic interval training. A protocol of total 5 weeks. Three sessions per week on alternate days will be done under the supervision of physiotherapist.
  All outcome measurements would be performed first at baseline and terminal after the 5 weeks intervention period
  Interventions: Other: interventional group A

INTERVENTIONS:
Other: Experimental Group — The interventional group will perform aerobic training (stationary cycling) 3 days a week for 5 weeks, starting with 40-60% heart rate reserve (HRR) for 20-30 minutes, with thein the first week and increasing to 40-85% HRR, maintaining a target heart rate of 40-60% HRR at the lower end and 75-85% HRR at the upper end, following a 1:4 work-to-rest ratio for 30-40 minutes in subsequent weeks, with the warm up of 5 mins before the session and a cool down of 5-7 mins after every seasion. Exercise heart rate will be calculated using the Karvonen formula for the base line week and the following weeks.Following each aerobic session, they'll practice Alternate Nostril Breathing (ANB), beginning with 5 minutes in the first week and progressing to 10 minutes thereafter. ANB involves specific hand positioning and breathing techniques to promote relaxation and balance. All sessions will be supervised by a physiotherapist.
  Arms: Interventional group (Group B)
Other: interventional group A — In interventional group 'A' participants will perform aerobic training for 3 days a week for 30-40 minutes a day for 5 consecutive weeks. Exercise heart rate will be calculated using the Karvonen formula. For the first base line week the aerobic session begins with a 5-minute warm-up. The primary cardiovascular component involves using a cycle ergometer (stationary cycling) at an intensity of 40-60% heart rate reserve (HRR) for 20-30 minutes. Finally, the workout will concludes with a cool-down phase lasting 5-7 minutes, allowing the heart rate to gradually return to baseline and preventing post-exercise hypotension. From the second week onwards, the aerobic training session will begin with a 5-minute warm-up to prepare the body and gradually increase heart rate. The main workout involves a cycle ergometer, maintaining a target heart rate of 40-60% HRR at the lower end and 75-85% HRR at the upper end, following a 1:4 work-to-rest ratio for 30-40 minutes. The session ends with a 5-7 min
  Arms: Interventional group (Group A)

SUMMARY:
Hypertension (HTN) is the foremost preventable risk factor for cardiovascular disease (CVD) and all-cause mortality, contributing to over 7 million deaths annually within the nearly 17 million attributed to CVD. Effective management through lifestyle modifications, including aerobic exercises specifically interval training presents a promising avenue for blood pressure regulation by promoting vasodilation and regulating the autonomic nervous system. Likewise, alternate nostril breathing has demonstrated efficacy in lowering blood pressure by optimizing oxygenation and improving endothelial function but their combined effect on BP measures is yet to be determined. Hence this study aims to determine the combined effects of aerobic interval training with and without alternate nostril breathing on blood pressure, rate pressure product and quality of life in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25- 50 years -males and females
* Patients diagnosed with stage 1 hypertension 130 - 139 / 80 - 89 mmHg and stage 2 hypertension, BP level ≥140/90 mmHg. according to AHA/ACC 2017 Guidelines-Individuals who are able to understand and follow the instructions for exercise

Exclusion Criteria:

* Diagnosed with any current infections
* subjects with diagnosed musculoskeletal or neurological conditions which hinder participation in physical activity program
* Active Smokers
* Those with any contraindication to exercise testing or training.
* Pregnant females

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
heart rate | 05 weeks
  heart rate will be measured by pulse oximeter
blood pressure | 05 weeks
  it will be measured by pulse oximeter
Rate pressure product | 05 weeks
  it will be evaluated by formula : systolic blood pressure x heart rate resting by using sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, 44000, Rawalpindi, Pakistan